CLINICAL TRIAL: NCT05153720
Title: Comparison of Ultrasound Guided Erector Spinae Block and Ultrasound Guided Caudal for Perioperative Analgesia in Pediatric Cancer Patients Undergoing Nephrectomy Surgeries: a Randomized Controlled Study
Brief Title: Erector Spinae Block Versus Caudal Block for Perioperative Analgesia in Pediatric Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Assistant Professor of Anesthesia and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AP2109-30109
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound guided erector spinae plane block (Experimental): Unilateral erector spinae plane block will be performed under ultrasound guidance
  Interventions: Procedure: Erector spinae plane block
- Ultrasound guided caudal block (Active Comparator): Caudal block will be formed under ultrasound guidance
  Interventions: Procedure: Caudal block

INTERVENTIONS:
Procedure: Erector spinae plane block — Ultrasound guided erector spinae plane block
  Arms: Ultrasound guided erector spinae plane block
Procedure: Caudal block — Ultrasound guided caudal block
  Arms: Ultrasound guided caudal block

SUMMARY:
The study aim to compare ultrasound guided erector spinae plane block versus ultrasound guided caudal block in perioperative analgesia for pediatric cancer patients

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Age >1 and <12
* patients undergoing nephrectomy surgeries

Exclusion Criteria:

* patients parental refusal
* local infection at the puncture site
* coagulopathy with INR> 1.6
* unstable cardiovascular disease
* patients allergic to medication used
* development or mental delay
* impaired liver and renal functions

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
opioid consumption | First 24 hours postoperatively
  postoperative morphine consumption

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Assistant Professor of Anesthesia and Pain Management, National Cancer Institute, Cairo University; Yasmen F Abdelghani, M.Sc, Principal Investigator — Assistant Lecturer of Anesthesia and Pain Management, National Cancer Institute, Cairo University
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided